CLINICAL TRIAL: NCT01312701
Title: Observational Immunomonitoring Study of NK/T and Myelocites Status in Cancer Patients and Controls
Brief Title: Study of Blood Immune Cells in Cancer Patients Compared to Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Hovav Nechushtan senior Lecturer MD PhD, Hadassah Hebrew University Medical center
Other Study IDs: zeta-im-1
Record Dates: First submitted 2011-03-01; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Solid Carcinoma
Keywords: cancer; immunomonitoring; CD247 -zeta chain; chronic inflamation; anticancertherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators will collect peripheral blood for facts analysis of intracellular levels of proteins.
  Some of these cells may be frozen for longer periods of time for comparison with other new samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cancer patients: as described patietns with solid cancer about to be treated with anticancer therapies
- control group: normal populations who domated blood for further use

SUMMARY:
Tumors have a systemic immune modifying effect. They affect the immune system similarly to states of chronic inflammation and these effects can:

* be monitored through analysis of nk t and myeloid cells mainly through studies of the zeta chain but also through other means
* may be decreased following effective anticancer therapy - may even be used to study the effectiveness of anticancer therapy
* are important to monitor if the investigators plan on formulation of systemic immune therapy Thus immumonitoring of systemic blood cells may turn out to be an important prognostic and predictive factor in many cancer types

DETAILED DESCRIPTION:
CD247 Known also as the zeta chain is important for relaying T-cell induced signal transduction.

Interestingly studies by Baniash and others have demonstrated that this chain is down regulated in states of chronic inflammation and cancer in peripheral blood T cells and also in NK cells However there has not been a prospective study of this marker in cancer and control patients such a study will reveal not only the levels of CD247 in immune cells of cancer patients compared to controls but may reveal the effect of anticancer therapies on CD247 in cancer patients such a study may contribute significantly to our ability to monitor systemic immune system characteristics in cancer patients and help in any further studies of immunomodulation such as vaccination schemes in such patients

ELIGIBILITY:
Inclusion Criteria:

* patients with cancer or blood donators agreeing to participate in the trial

Exclusion Criteria:

* other disease states which may cause chronic inflammation

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: controls - patients who were deemed eligible for blood donation cancer patients - patients with solid tumors who agreed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
changes in immune markers mainly cd247-zeta chain - levels in cancer patients undergoing therapy | 4-2013 24 month
  Hopefully by this time the investigators will be able to see if there are lower zeta chain intracellular expression levels in cancer patients and whether response to therapy enhances recovery of zeta chain
levels of zeta chain -cd247 in cancer patients | till begining of 2013 ( putative)
  intracellular levels of cd247 compared to other intracellular proteins and other markers of immune response will be monitored in patients with cancer and a control group in cancer patients the investigators will conduct several tests to analyze effects of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hovav Nechushtan, MD PhD, Principal Investigator — Oncology Dept Hadassah Hebrew University Medical Center
Locations (1):
- Oncology day care Oncology Dept Sharett Inst Hadassah Ein Kerem, Jerusalem, Israel

REFERENCES:
- [Background] Ezernitchi AV, Vaknin I, Cohen-Daniel L, Levy O, Manaster E, Halabi A, Pikarsky E, Shapira L, Baniyash M. TCR zeta down-regulation under chronic inflammation is mediated by myeloid suppressor cells differentially distributed between various lymphatic organs. J Immunol. 2006 Oct 1;177(7):4763-72. doi: 10.4049/jimmunol.177.7.4763. PMID 16982917